CLINICAL TRIAL: NCT05055518
Title: Phase I Study on Safety, Tolerance, and Pharmacokinetics of APL-102 Capsule in Patients With Advanced Solid Tumors
Brief Title: APL-102 Capsule in Patients With Advanced Solid Tumors
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Voluntarily suspended (due to adjustments in corporate development strategy, not for reasons related to safety or efficacy.)
Sponsor: Apollomics Inc. (Industry)
Collaborators: Zhejiang CrownMab Biotech Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL-102-01
Record Dates: First submitted 2021-08-22; First posted 2021-09-24 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to a dose level of APL-102 in the order of study entry. A total of seven therapeutic dose levels (1mg, 2mg, 3mg, 5mg, 7mg, 9mg and 11mg) are planned. To reduce the number of subjects exposed to potentially ineffective doses and protect the rights and interests of subjects, rapid titration was used in the low-dose group (1 mg, 2 mg, 3 mg); When approaching the expected effective dose of 5 mg, the "3 + 3" study design was used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A Phase I, open-labeled multicenter study (Experimental): APL-102 Capsules
  Interventions: Drug: APL-102 Capsules

INTERVENTIONS:
Drug: APL-102 Capsules — Dose escalation: A total of seven dose levels (1mg, 2mg, 3mg, 5mg, 7mg, 9mg and 11mg) are planned.
  Dose extension: After RP2D determined, the RP2D dose level will be extended to enroll 6-10 subjects to further evaluated the safety and antitumor activity of APL-102.
  Other Names: No other name so far

SUMMARY:
This study will evaluate the safety and tolerability of APL-102 Capsule and characterize the pharmacokinetic (PK) profile in advanced solid tumor patients.

DETAILED DESCRIPTION:
This study is an open, multicenter dose-escalation study to evaluate the safety and tolerance of APL-102 and obtain the relevant data of APL-102 in patients with advanced solid tumors. In the dose escalation stage, based on the incidence of dose limited toxicity (DLT) and adverse event (AE), explore and determine the maximum tolerated dose (MTD) and phase II recommended dose (RP2D). After RP2D and administration protocol are determined, an extended study will be conducted on 6-10 subjects to further evaluate the safety and antitumor activity of APL-102.

ELIGIBILITY:
Major Inclusion Criteria:

1. Male or female, age ≥ 18 and ≤ 75 years old.
2. Patients with unresectable or metastatic advanced solid tumors confirmed by histology or cytology, and after the failure of standard treatment, or cannot tolerate standard treatment, or have no standard treatment.
3. There were measurable lesions according to the efficacy evaluation criteria of solid tumors (RECIST version 1.1).
4. Eastern Cooperative Oncology Group(ECOG) performance status score is 0 to 1.
5. Life expectancy is more than 3 months after the first administration.
6. The organ function level must meet the following requirements:

   Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.0× upper limit of normal value (ULN) (patients with liver metastasis≤ 5 × ULN). Serum bilirubin ≤ 1.5×ULN (total bilirubin ≤ 3×ULN in patients with Gilbert syndrome). Absolute neutrophil count ≥ 1.5×10^9/L. Platelet count ≥ 100×10^9/ L. Hemoglobin ≥ 9 g / dL.
7. No other chemotherapy was received within four weeks before the first administration of the trial; All previous anti-tumor treatments, including targeted therapy and endocrine therapy, shall pass through at least five half-lives (or no more than 28 days) after receiving targeted therapy/endocrine therapy, and patient shall recover to the standard level specified in the test from the toxic reaction of the treatment.
8. For patients who have received radiotherapy for spine and/or peripheral limbs, they can only be enrolled after four weeks and two weeks before the first administration and should recover from the toxic reaction of treatment to the standard level specified in the study.
9. No major surgery was performed within four weeks before the first administration of APL-102., etc.

Major Exclusion Criteria:

1. In addition to the malignancies in the study, patients with systemic diseases leading to poor medical risk (such as uncontrollable infection in the active phase).
2. Life-threatening diseases, severe organ dysfunction, interference with the absorption or metabolism of APL-102, or other reasons that the researchers believe may endanger the safety of subjects or affect the integrity of research results.
3. Patients with a history of heart disease or potential risk of heart disease.
4. Patients with low circulatory function as defined by the New York Heart Association's (NYHA) functional criteria.
5. Patients with a definite diagnosis of chronic obstructive pulmonary disease, bronchial asthma or interstitial lung disease, or patients with forced expiratory volume in one second/ forced vital capacity (FEV1/FVC) ratio < 70% in pulmonary function test.
6. Patients with decompensated cirrhosis or history of allogeneic bone marrow transplantation or organ transplantation.
7. Patients in repeated resting states during screening had mean systolic blood pressure ≥140 mmHg, diastolic blood pressure ≥90 mmHg, or positive proteinuria (allowing antihypertensive agents to control blood pressure).
8. Have a history of human immunodeficiency virus (HIV) infection or HIV antibody positive; or seropositive results consistent with active infection for hepatitis B virus (in case of only hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive, the examination of Hepatitis B (HBV) DNA copy number is needed: HBV DNA copy number must not exceed 1,000 copies/mL or 200 IU/mL.) or hepatitis C virus.
9. Patients with the symptomatic primary brain tumor and/or secondary brain metastasis, uncontrollable antiepileptic drugs and requiring high-dose steroid treatment. Or cerebrovascular accident, transient ischemic attack, or intermittent claudication within six months before treatment.
10. Pregnant or lactating patients., etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
DLT | 36 days
  Dose limiting toxicities
Adverse Events (AEs) | From time of informed consent signature to 30 days after the subject's last visit (approximately 1 year)
  Adverse events occurred in all subjects during the study treatment according to the National Cancer Institute Common Terminology Standard for adverse events (NCI CTCAE) standard version 5.0

SECONDARY OUTCOMES:
Incidence of Adverse Events | From time of informed consent signature to 30 days after the subject's last visit (approximately 1 year)
  The incidence of all adverse events with different severity (NCI CTCAE 5.0)
Objective response rate(ORR) | Approximately 1 year
  The objective response rate in patients of advanced solid tumors
Duration of response(DOR) | Approximately 1 year
  The duration of response in patients of advanced solid tumors
Progression-free survival(PFS) | Approximately 1 year
  The progression-free survival in patients of advanced solid tumors
Overall survival(OS) | Approximately 1 year
  The overall survival in patients of advanced solid tumors
Peak plasma concentration (Cmax) | 36 days
  To assess the pharmacokinetic profile in patients with advanced solid tumors.
Time to reach Cmax (Tmax) | 36 days
  To assess the pharmacokinetic profile in patients with advanced solid tumors.
The area under the plasma concentration-time curve from time zero to the last measurable time point (AUC0-t) | 36 days
  To assess the pharmacokinetic profile in patients with advanced solid tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Yihebali Chi, PhD, Principal Investigator — Investigator
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No